CLINICAL TRIAL: NCT05777473
Title: Tipping Point: Using Social Network Theory to Accelerate Scale and Impact
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Save the Children (Other)
Responsible Party: Principal Investigator, Jay G. Silverman, PhD, Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 201921
Record Dates: First submitted 2023-02-22; First posted 2023-03-21 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Contraception
Keywords: Contraception Behavior; Female Adolescent; Married; West Africa; Family Planning; Contraceptive Use; Birth Spacing
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Intervention Model Description: Three-arm cluster randomized controlled trial (cRCT)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kulawa (Experimental): This arm will receive the standard Kulawa intervention. Kulawa is a USAID-funded program that seeks to change FP-related behaviors among young, low parity women at scale in Niger. Kulawa, implemented by Save the Children U.S. aims to increase use of quality FP services of all WRA, including young women ages 15-24 years, in 15 districts of Niger across 3 regions (Tillaberi, Maradi, and Zinder), covering a population of 12.5 million. Kulawa will address individual, social, and health system constraints to FP use through interventions to change behavior and influence social norms that govern FP use and related gender outcomes as well as interventions to improve FP service availability and quality. Kulawa SBC programming at the community-level will include small groups for young, low parity women and girls (ages 15-24) and community dialogues.
  Interventions: Behavioral: Household Visits; Behavioral: Small Groups
- Kulawa SN (Tipping Point) (Experimental): This arm will receive the Kulawa intervention, with a social network-informed intervention (KulawaSN) layered on top. In this arm 50% of eligible women will be paired with an alter to receive the adapted intervention. The social network intervention will involve pairing up young married adolescents and women with someone identified as influential in their social networks and enrolling them in the Kulawa FP programming together.
  Interventions: Behavioral: Household Visits; Behavioral: Small Groups; Behavioral: Adopt-a-Friend
- Control (No Intervention): This arm will serve as the control condition. Individuals in these villages will receive neither intervention (including any other FP-relevant SBC program)

INTERVENTIONS:
Behavioral: Household Visits — Household visits will be conducted to build trust in the health system, educate regarding different forms of modern contraception, (how administered, how they work, availability), dispel related myths (i.e., those regarding infertility), promote the health advantages of birth spacing, and create related dialogue among adolescent wives and other household members present during these visits. The community health worker will provide and resupply oral contraceptive pills and condoms to interested participants and will accompany the married adolescent to the nearest health facility for other forms of contraception, if requested to do so. To complement the household visits to married female adolescents, male community health workers will conduct home visits to discuss healthy timing and spacing of pregnancy with husbands of adolescent females, provide education on different forms of contraception, and discuss concerns husbands may have regarding use of contraception.
  Arms: Kulawa; Kulawa SN (Tipping Point)
Behavioral: Small Groups — In the wife-only groups, adolescent wives will be convened by trained adult female community members to learn and discuss a broad range of gender and health-related topics, with a focus on modern contraception, and cultivate self-efficacy, social support and life skills. The small groups will be led by trained female small group mentors who are trained peers and will follow a designated curriculum consisting of different topics each week. The husband groups will focus on fostering reflection and dialogue to contribute to more equitable gender norms, support for contraception use for HTSP, positive health seeking behavior for them and their families, and increased couples communication and joint SRH decision-making.
  Arms: Kulawa; Kulawa SN (Tipping Point)
Behavioral: Adopt-a-Friend — The "Adopt a Friend" approach aims to promote the dissemination and discussion of new information and ideas among peers who are not directly involved in program activities. This involves asking each participant to choose a friend with whom she will share what she learns in home visits and her reflections. Adolescent girls will support each other in seeking sexual and reproductive health information or services if needed.
  Arms: Kulawa SN (Tipping Point)

SUMMARY:
This study will assess the nature and impact of social norms and networks to promote FP (Family Planning) intervention effects among low parity, married adolescent and young women in the Maradi region of Niger. Research activities will be layered on top of the USAID-funded Kulawa FP program that seeks to change FP-related behaviors among young, low parity women at scale in Niger in a subset of implementing villages. Kulawa, implemented by Save the Children U.S. (SCUS) and funded by USAID (2020-2025), will include small-group discussion for young, low parity girls coupled with community dialogues to address individual, social, and health system constraints to FP use and influence social norms that govern FP use. UCSD will not provide any services or implement any interventions as part of this study.

DETAILED DESCRIPTION:
Research Design: The investigators will use a three-arm cluster randomized controlled trial (cRCT) to determine the effectiveness and scalability of a social network approach to increasing knowledge and uptake of family planning in low-parity, married adolescent and young women aged 15 to 24. This study will take place across 51 randomly selected villages in the Maradi region of Niger from the districts of Aguie, Gazaoua, and Tessauoua. Approximately 450 villages exist across these three districts, of which 302 meet our eligibility criteria. Eligibility criteria for selection of villages includes villages being 1) located in the Aguie, Gazaoua, or Tessauoua), 2) rural (i.e., not designated as a market town or city), 3) Hausa or Zarma-speaking, 4) total population size of the village consistent with a population of approximately 30 married adolescent girls, and 5) located within 5 km of a health clinic (i.e., centre de santé intégré). Once selected, villages will be randomized to one of three treatment arms (17 villages/arm). Depending on the arm, low parity, married adolescent and young women will receive either the standard Kulawa program (Arm 1), the Kulawa program adapted with a social network approach (Arm 2), or no FP programming (Arm 3, i.e., control). The Kulawa program adapted with a social network approach will be developed by Save the Children based on formative research and will include delivery to both female participants and one of their female alters (a nominated socially connected community member). Note that in villages selected for Arm 2, 50% of eligible participants will be randomly selected to receive the Kulawa intervention with the social network approach, to test effects of diffusion and accelerated impact. The other 50% of eligible participants in Arm 2 will receive the program, if successful, after 24 months (see below and Table 1 for details of participants).

Formative Research: The investigators will begin by collecting data for formative research and intervention development. This research will involve conducting qualitative social network interviews villages proximal to those in the treatment arm. Research aims will be to understand the best way to develop the social network intervention modification, including developing methods for identifying alters to include in the Kulawa social network intervention. Qualitative interviews will also help the investigators measure norm and behavior change among this population. Approximately 20 interviews will be conducted, 10 interviews with low parity, married adolescent and young women ages 15-24 years and 10 interviews with an influential individual that they name (female member of the community, minimum age 15 years). Each interview will take 45-60 minutes. Interviews will be audio recorded, translated, and transcribed.

Pilot: Survey assessments will include FP use and related behaviors, decision-making, personal attitudes, social norms, and social network influences. Surveys will be piloted in two villages comparable to those selected for the trial, among eligible female participants (approx. 30 per village), their nominated alters, and husbands. Based on findings, the study tools and social network intervention strategy will be refined.

Effectiveness Evaluation: The 3-arm RCT trial will take place across 51 villages (i.e., 17 villages per district) in the Maradi region of Niger randomly assigned to 1 of the 3 treatment arms. Within each village, households with eligible, married females (see Human subjects for eligibility criteria) will be enumerated by village elders. All eligible females in the villages (approx. 30/village) will be approached for recruitment (see Recruitment for details). The study will have three longitudinal waves of data collection: baseline (conducted immediately prior to the intervention), midline (conducted 12-months post the start of intervention implementation) and an endline (conducted 24-months post the start of intervention implementation). Survey interviews will be conducted with all eligible low parity, married adolescent and young women in each village (N=1530, 510 each arm, see human subjects for eligibility criteria) and take 45-60 minutes. Surveys will be conducted by a trained research assistant orally in Hausa or Zarma (at the participants choosing) who will record participant responses on a tablet computer. At each time point, participating low parity, married adolescent and young women (egos) will name a female influential to her FP decision-making (an alter) using the same approach described in the Preliminary studies. This individual (known as the first-degree alter) will also be interviewed at each time point in the same fashion as the original respondent (1530 per wave). These individuals will also nominate another influential individual (known as the second-degree alter). In treatment Arms 1 & 2 only, the second-degree alters will also be interviewed in the same fashion (N=1020 per wave). Second-degree alters will not be interviewed in control villages. If individuals are named by multiple participants, they will not be re-interviewed. In treatment Arms 1 & 2 only, husbands of originally recruited participants will also be surveyed (N=1020) via a verbal 45-60-minute survey interview.

Analysis & Dissemination: Difference-in-differences models will be used to detect the differences between baseline and follow-up across different arms. Geographic analysis will also be conducted to test for the effect of geographic factors on behavior and norm adoption. Data will be disseminated after each wave of data collection to local, national, regional, and global stakeholders.

ELIGIBILITY:
Inclusion Criteria:

For Women:

* Married
* 15-24 years old; or mother-in-law of married adolescent (or replacement MIL)
* Residing in the village where recruitment is taking place
* Providing informed consent

For Men:

* Must be the husband to an eligible adolescent participating in the study
* Providing informed consent

Exclusion Criteria:

-

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 3825 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Contraception Use Questionnaire (individual items, not a scale) | Baseline, 12-month Midline, and 24-month Endline
  Change in use of effective methods of contraception
Intentions To Use Contraception Questionnaire (individual items, not a scale) | Baseline, 12-month Midline, and 24-month Endline
  Change in behavioral intentions regarding effective contraceptive use

SECONDARY OUTCOMES:
Social Norms regarding gender equity Questionnaire (individual items, not a scale) | Baseline, 12-month Midline, and 24-month Endline
  Change in social norms regarding husbands physical and sexual violence toward wives, women's autonomy and husbands control related to family life
Female Empowerment Questionnaire (individual items, not a scale) | Baseline, 12-month Midline, and 24-month Endline
  Change in autonomy, decision-making, freedom from violence and control, especially with regard to contraceptive use
Acceptance of effective contraceptive methods Questionnaire (individual items, not a scale) | Baseline, 12-month Midline, and 24-month Endline
  Change in attitudes and beliefs regarding use of contraceptive methods for birth spacing

CONTACTS AND LOCATIONS:
Locations (1):
- Center on Gender Equity and Health, University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No